CLINICAL TRIAL: NCT02447575
Title: Detecting Errors In Using Metered Dose Inhalers (MDI) Among Asthma And Chronic Obstructive Pulmonary Disease (COPD) Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: William Marsh Rice University (Other)
Responsible Party: Principal Investigator, Nicola Hanania, Associate Professor of Medicine, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: H36079
Record Dates: First submitted 2015-05-12; First posted 2015-05-19 (Estimated); Results first posted 2020-10-09 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-09

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MDI use Evaluation (Other): All subjects took 2 or more puffs of the placebo metered dose inhaler (MDI), attaching the Cognita electronic flowmeter to show measurements during the MDI use.
  The inhaler technique is also evaluated by study staff prior to an education demonstration.
  Interventions: Other: Education on Use of MDI

INTERVENTIONS:
Other: Education on Use of MDI — After the subject demonstrated the use of MDI with the electronic flowmeter in place, the intervention was provided- a short verbal education to demonstrate the correct use of MDI.

SUMMARY:
Metered Dose Inhaler (MDI) and Dry Powdered Inhaler (DPI) are the two most common devices used to deliver medicine in conditions such as asthma and chronic obstructive pulmonary disease. It is well-known that most patients do not use correct technique when using a metered dose inhaler. This leads to poor control of their disease. This study is being done so the investigators can record the patient using the metered dose inhaler before and after a short teaching session. This information will be fed into an invitro system (device) to allow the researchers to study the effect of error on drug delivery. The device being used is the Rice R3 electronic flowmeter.

DETAILED DESCRIPTION:
Metered Dose Inhaler (MDI) and Dry Powdered Inhaler (DPI) are the two most common platforms to deliver medicine for patients suffering from Asthma and chronic obstructive pulmonary disease, and are used for dispensing both controller and rescue medications. Despite well-known methods to manage Asthma and COPD, nearly 70-90% of the patients do not display correct technique in using an inhaler. Poor management and control of the disease due to inadequate inhaler usage has resulted in rising rates of hospitalizations, making chronic respiratory diseases among the top five causes of death worldwide. Through this study we aim to record the technique of MDI usage among Asthma and COPD patient and understand the errors in their technique. The various parameters of inhaler usage where patients can make an error are 1. Tidal volume, 2. inspiration flow rate, 3. Inspiration flow volume, 4. Timing of actuation of inhaler and 5. Breath-holding. The parameters will be recorded by the Cognita R3 electronic flowmeter for each patient and the errors in each MDI usage will be noted. Using ex-vivo modelling, the patient's MDI technique recorded will be used to study the impact of errors in technique on efficiency of MDI drug delivery.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a physician diagnosis of asthma or COPD taking inhaled medications using MDI
* Age >18 years
* Able to read and sign consent document

Exclusion Criteria:

* Patients having acute exacerbation
* Patients who are unable to take medication from an MDI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-02; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola A Hanania, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Biswas R, Hanania NA, Sabharwal A. Factors Determining In Vitro Lung Deposition of Albuterol Aerosol Delivered by Ventolin Metered-Dose Inhaler. J Aerosol Med Pulm Drug Deliv. 2017 Aug;30(4):256-266. doi: 10.1089/jamp.2015.1278. Epub 2017 Feb 3. PMID 28157430

RESULTS

PARTICIPANT FLOW:
Groups:
- MDI Use Evaluation: Patients perform metered dose inhaler (MDI) technique, attaching the Cognita electronic flowmeter to show measurements during the MDI use. These are evaluated by study staff prior to an education demonstration. The intervention is a short educational presentation on the correct use of the MDI.
  MDI use Evaluation: Subject will demonstrate the use of MDI) with an electronic flowmeter in place before a short education process to demonstrate current use of MDI
Period: Overall Study
Arm/Group | MDI Use Evaluation
Started | 23 (23 subjects were enrolled in the study: http://dx.doi.org/10.1016/j.chest.2016.08.017)
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 23 physician-diagnosed Asthma/COPD patients were recruited for the study.
Groups:
- MDI Use Evaluation: This was a single-arm study. All participants were instructed to use the MDI with the flow meter to gauge the correctness of use.
Arm/Group | MDI Use Evaluation
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.65 (13.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Inhaler Use Correctness
Description: This is an observational study, the aim is to record a variety of MDI usage techniques performed by patients. The technique is scored out of 7 for the following 7 steps:
  1. Shaking (0 = not shaken, 1 = shaken)
  2. Coordination (0 = MDI actuated before inhalation start, 1 = MDI actuated after inhalation start)
  3. Flow rate (0 = mean inspiratory flow rate <30L/min or greater than 60L/min, 1 = mean inspiratory flow rate between 30-60L/min)
  4. Duration of inhalation (0 = duration of inhalation <3 sec, 1 = duration of inhalation >=3sec)
  5. Orientation of inhaler (0 = inhaler not upright = > 30° from the vertical position, 1 = inhaler upright = within 30° from the vertical position)
  6. Number of exhalation (0 = exhalation during inhaler use, 1 = no exhalations)
  7. Single Actuation (0 = less than 0 or more than 1 inhaler actuation, 1 = exactly 1 inhaler actuation)
  The total score is a minimum of 0 correct steps if all the steps are incorrect to a maximum of 7 correct steps.
Time Frame: Single event- Outcome measured per inhaler puff, during the single clinic visit.
Population: 23 subjects completed the study.
  Partial results were published in:
  1. Biswas, Rajoshi et al., Journal of aerosol medicine and pulmonary drug delivery 30.4 (2017): 256-266.
  Complete results were published in:
  1. Biswas, Rajoshi, et al., Chest Journal 150.4_S (2016).
Measure: Mean (Standard Deviation); unit: correct steps
Arm/Group | MDI Use Evaluation
Number analyzed (Participants) | 23
correct steps | 3.52 (1.25)

ADVERSE EVENTS:
Time Frame: 1 day.
Description: The study was a single inhaler use event with placebo medication. The risk of adverse events with less than 4 doses of placebo medication is low. The reporting is based on self-report by the participant on the day of the placebo MDI use. The event is reported if a participant faced and reported an adverse event post MDI use at the clinic/study visit on the day of the study visit.
Groups:
- Single Arm Study I: This was a single-arm study. All participants were instructed to use the MDI with the flow meter to gauge the correctness of use.
Arm/Group | Single Arm Study I
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT02447575/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/75/NCT02447575/ICF_001.pdf